CLINICAL TRIAL: NCT00005594
Title: Phase II Trial of ISIS 2503, an Antisense Inhibitor of H-Ras, in Patients With Advanced Pancreatic Cancer
Brief Title: ISIS 2503 in Treating Patients With Advanced Cancer of the Pancreas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: James Posey, MD/ Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067701; UAB-9915 (Other Grant/Funding Number: 0001215); ISIS-2503-CS5; UAB-F990526011; NCI-G00-1730
Record Dates: First submitted 2000-05-02; First posted 2004-05-03 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2010-12

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — ISIS 2503

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ISIS 2503 (Experimental): All patients will begin treatment at a dose of 6 mg/kg/day of ISIS 2503. ISIS 2503 at the assigned dose will be given as a continuous i.v. infusion over the first 14 days of a 21-day treatment cycle. No drug will be administered during the third week of each treatment cycle.
  Interventions: Drug: ISIS 2503

INTERVENTIONS:
Drug: ISIS 2503 — Beginning dosage of ISIS 2503 is 6 mg/kg/day given as a continuous i.v. infusion over the first 14 days of a 21-day treatment cycle. This will be repeated for the first two weeks of every three-week treatment cycle.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of ISIS 2503 in treating patients who have advanced cancer of the pancreas.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate and time to progression in patients with advanced adenocarcinoma of the pancreas who are treated with ISIS 2503. II. Determine the duration of response in these patients receiving this regimen. III. Characterize the safety profile of ISIS 2503 at the recommended phase II dose and schedule in these patients.

OUTLINE: Patients receive ISIS 2503 IV continuously for 14 days. Treatment continues every 21 days for a minimum of 3 courses in the absence of unacceptable toxicity or disease progression.

PROJECTED ACCRUAL: A total of 14-27 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced adenocarcinoma of the pancreas that is considered inoperable Measurable disease with at least 1 lesion measuring at least 2 cm in widest diameter identifiable on CT or MRI scan

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count greater than 1,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL Renal: Creatinine no greater than 2.0 mg/dL Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective barrier contraception during and for 6 months after study No underlying disease state associated with active bleeding No active infection requiring therapy No other prior malignancy within the past 5 years except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent biologic therapy for pancreatic cancer Chemotherapy: No prior chemotherapy for pancreatic cancer except for fluorouracil and/or gemcitabine administered as a radiosensitizer No other concurrent chemotherapy for pancreatic cancer Endocrine therapy: Not specified Radiotherapy: Prior radiotherapy allowed provided indicator lesions not within prior radiation port Recovered from toxicity No concurrent radiotherapy for pancreatic cancer Surgery: See Disease Characteristics Other: No concurrent anticoagulation therapy with heparin No other concurrent approved or experimental cancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2000-07; Primary Completion 2000-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure of this study is to estimate the response rate and observe the time to tumor progression of the patients treated on this study. | 24 weeks

SECONDARY OUTCOMES:
Determine the duration of response in responding patients. Further characterize the safety profile of ISIS 2503 at the recommended dose and schedule. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James A. Posey, MD, Study Chair — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Norris Cotton Cancer Center, Lebanon, New Hampshire